CLINICAL TRIAL: NCT04443985
Title: A Cohort of Predictive Factor of Pathologic Complete Response After Preoperative Neoadjuvant in Rectum Cancer
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: Ramathibodi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MURA2019/249
Record Dates: First submitted 2020-06-11; First posted 2020-06-23 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Rectum Cancer
Keywords: Preoperative chemoradiation; Rectum cancer; Pathological complete response
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Due to colorectal cancer is the fourth most common malignancy in the world. Some patients had present locally advance stage and need to preoperative concurrent chemoradiation (CCRT) before radical surgery. But predictor for pathologic complete response (pCR) after preoperative CCRT remain unclear.

Objectives: To identify possible factor for predict of pCR of rectal cancer after preoperative CCRT.

DETAILED DESCRIPTION:
After permission was obtained from our institutional review board, a cohort of patients who were diagnosed with rectal cancer and received chemoradiation between January 2011 to December 2017 at Ramathibodi hospital, Bangkok were analyzed. Patients who were not received neoadjuvant chemoradiation therapy, loss follow-up, incomplete data in the record, distant organ metastasis and who was not received colorectal surgery were excluded as study flow diagram. Age, sex, performance status, smoking, initial Hb level (g/mL), CEA level (ng/dL), distance of tumor from anal verge, diagnostic variables, clinical T staging, preoperative thickness and length from computer tomography scan (CT scan), organ metastasis before treatment, histology, treatment course, and outcomes after treatment were collected and analyzed.Total dose of radiation, interval time from CCRT to operation, and chemotherapy regimens were also collected between and after treatment. After preoperative CCRT, the radical rectal surgery was performed by eight experienced general surgeons and surgical oncologist using open and laparoscopic techniques. Perioperative data were collected and histology was evaluated by an experienced pathologists. For pathological classification, pathological responses were divided in 2 groups i.e., pathologic complete response (pCR group) and non-pCR group, (partial response, stable disease, and disease progression). Margin of lesions were classified as proximal, distal and circumferential margins. Lymph nodes status after surgery were specified as total lymph nodes harvested and positive lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* rectal cancer and received preoperative chemoradiation

Exclusion Criteria:

* distant organ metastasis
* previous colorectal surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with rectal cancer and received chemoradiation
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Stage | 1 month
  Pathological of Tumor follow by The American Joint Committee on Cancer (AJCC) edition 8
Lymph node | 1 month
  Pathological of lymph node follow by The American Joint Committee on Cancer (AJCC) edition 8

CONTACTS AND LOCATIONS:
Overall Officials: Chairat Supsamutchai, MD, Study Chair — Ramathibodi Hospital, Mahidol University
Locations (1):
- Chairat Supsamutchai, Bangkok, Bankok, Thailand

IPD SHARING:
Plan to Share IPD: No